CLINICAL TRIAL: NCT06020261
Title: The Efficacy of Parent Management Training to Treat Irritability
Brief Title: Parent Management Training to Treat Irritability
Acronym: PMT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-0065
Record Dates: First submitted 2023-08-25; First posted 2023-08-31 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Irritable Mood; Temper Tantrum; Anger
Keywords: irritability; anger; parenting; temper outbursts; Parent Management Training
MeSH Terms: interventions — Behavior Therapy

STUDY DESIGN:
Intervention Model Description: All participants will receive 12 sessions of Parent Management Training to treat irritability. Participant children and their parents will complete pre-treatment, mid treatment, and post-treatment assessments to determine if there is any improvement in irritability or other areas of functioning.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Parent Management Training (Experimental): 12 sessions of manualized Parent Management Training for irritability developed by the National Institute of Mental Health.
  Interventions: Behavioral: Parent Management Training

INTERVENTIONS:
Behavioral: Parent Management Training — developing parenting skills and competencies dealing with oppositional and irritable behaviors in the child.
  Other Names: behavioral treatment

SUMMARY:
The goal of this clinical trial is to see if 12 sessions of a Parent Management Training program can treat irritability in children aged 10-14 years old. The main question it aims to answer are:

* Can a Parent Management Training for parents reduce anger outbursts and cranky moods in their children?
* Can Parent Management Training be done in an outpatient clinic and do parents like it?

Up to 18 families can join this study. This study will be used to set up a larger study in the Fall of 2025.

Parent participants will complete 12 sessions of Parent Management Training for Irritability. Each session will be 45-55 minutes weekly. They will also participate in the assessments of their child before, during and after treatment.

Child participants will do assessments before, during and after the Parent Management Training treatment.

DETAILED DESCRIPTION:
Up to 18 families will be consented for this Parent Management Training (PMT) to Treat Irritability study in order to meet the aim of having 12 families complete the study. The child and a parent will complete pre-treatment evaluations about the child's mental health, behavior and cognitive functioning. Participants who meet inclusion criteria (age 10-14 with significant irritability) and do not meet exclusion criteria (e.g. Autism, Bipolar disorder, active PTSD, serious medical issues or Intellectual disability) will be invited to join the trial. All participants will receive the 12 PMT sessions from a licensed mental health professional. The PMT sessions will focus on the parents only, but both the parent and child will complete standardized measures and interview with a clinician in the middle of the treatment. After the 12 sessions of PMT, the parent and child will complete a post-treatment assessment. Pre and post treatments assessments will be compared to determine changes in the child's irritability and other areas of functioning.

ELIGIBILITY:
Inclusion Criteria:

* clinically significant irritability (Clinician Affective Reactivity Index 30 or greater)
* parent or guardian willing to participate in treatment with the child

Exclusion Criteria:

* psychiatric instability (danger to self/others, risky substance abuse)
* current active Post-Traumatic Stress Disorder (PTSD) or a severe active stressor (e.g. child abuse)
* history of severe psychopathology with an established alternate treatment (e.g. autism spectrum disorder, bipolar disorder, schizophrenia, intellectual disability)
* general medical condition that may be driving irritability or prevent generalizable physiologic measures.
* screen positive for an intellectual disability via Wechsler Abbreviated Scale of Intelligence Second Edition (WASI II) estimated Intelligence Quotient (IQ)<70.

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2025-06-12 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Demonstrate the feasibility of Parent Management Training (PMT) procedures | 5 months
  The study team will implement a PMT protocol with fidelity and acceptability assessments. A member of the study team will complete independent fidelity ratings of 50% of recorded sessions using the Cognitive Behavior Therapy for Irritability Adherence Scale. The Working Alliance Inventory (WAI) (revised short form) will be used by the clinician and the parent to rate engagement in treatment after each PMT session. There are no established benchmarks for this measure, but it will provide information about the acceptability of the treatment by rating the alliance between the therapist and the parent.

SECONDARY OUTCOMES:
Change in irritability | 5 months
  Participants will report a decrease in irritability as measured by the Revised Affective Reactivity Index-Clinician (ARI-CL). The ARI-CL rates temper outbursts, irritable moods and impairment. Total scores range from 0-50, with a score over 30 indicating severe clinical irritability and lower scores indicating lower irritability.

CONTACTS AND LOCATIONS:
Overall Officials: Joel Stoddard, MD, Principal Investigator — University of Colorado Denver, Anschutz Medical Campus; Joel Stoddard, MD, Principal Investigator — University of Colorado Denver Anschutz
Locations (1):
- Childrens Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No